CLINICAL TRIAL: NCT06390748
Title: Investigating the Immunomodulatory Effects of Esmolol in Sepsis Management and Its Impact on Patient Outcomes
Brief Title: Esmolol in Sepsis Management:Evaluating Immunomodulatory Effects and Impact on Patient Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lin Chen (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, Professor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SichuanPPHLC02
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Sepsis; Lymphocyte Disorder T; Immunologic Paralysis; Catecholamine; Overproduction; Beta-Blocker; Cytokine Storm; Sympathetic Nervous System Diseases
Keywords: Esmolol; Sepsis; Immune modulation; T-cell function; Inflammatory markers; Sympathetic Nervous System
MeSH Terms: conditions — Sepsis; Cytokine Release Syndrome; Autonomic Nervous System Diseases | interventions — esmolol

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment model to investigate the effects of Esmolol on patients with sepsis. Participants are randomly assigned to one of two groups. The first group, the intervention group, receives Esmolol in addition to the standard sepsis care, which includes antibiotics, fluid resuscitation, and other supportive therapies. Esmolol dosing is adjusted to achieve and maintain specific heart rate targets, and cardiac monitoring through daily electrocardiograms is implemented to track QT interval changes. The second group, the control group, receives only the standard sepsis care without any additional interventions.
Who Masked: Participant
Masking Description: This study employs a single-blind design where the participants are blinded to their treatment assignments. In this setup, the patients do not know whether they are receiving the intervention (Esmolol) or are in the control group receiving only standard sepsis care. This blinding is essential to mitigate placebo effects and bias in patient-reported outcomes. However, the care providers, as well as the investigators and outcomes assessors, are aware of the treatment assignments. This knowledge allows them to manage the care more effectively while maintaining a robust observational stance on the impact of the interventions. The single-blind design is chosen to ensure the integrity of the data collected, particularly in measuring clinical outcomes and patient responses, without influencing the patients' perceptions or expectations about the treatment they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care plus esmolol (Experimental): Patients in this group were administered Esmolol, a beta-1 selective adrenergic blocker, alongside the standard sepsis care protocols. The dosage of Esmolol was adjusted to maintain heart rate within predefined targets. Additionally, daily electrocardiogram (ECG) monitoring was conducted to assess changes in the QT interval, a critical measure given the potential cardiac effects of beta-blockers. This group aimed to explore not only the immunomodulatory effects of Esmolol but also its safety profile in terms of cardiac function in septic patients.
  Interventions: Drug: esmolol
- standard care (No Intervention): Patients in this cohort received the standard of care for sepsis without any additional intervention. This treatment included antibiotics, fluids, and other supportive therapies as dictated by current clinical guidelines for sepsis management.

INTERVENTIONS:
Drug: esmolol — The primary intervention is the administration of Esmolol. Esmolol was specifically used to evaluate its immunomodulatory effects in patients with sepsis in the study. The dosage was tailored to achieve optimal heart rate control, an integral part of the therapeutic strategy aiming to mitigate the hyperadrenergic state often seen in sepsis. Alongside Esmolol, daily electrocardiogram (ECG) monitoring was incorporated to observe any changes in the QT interval, ensuring cardiac safety due to the known potential cardiac effects of beta-blockers.
  Arms: standard care plus esmolol

SUMMARY:
Evaluate the effectiveness of esmolol, a selective β1-adrenergic receptor blocker, in modulating immune responses and improving patient outcomes in sepsis.

DETAILED DESCRIPTION:
The research aimed to investigate the immunomodulatory effects of Esmolol in sepsis treatment. A comprehensive study was conducted, incorporating both direct experimental assays and data extraction from Electronic Health Records (EHR) to evaluate physiological and immunological responses in septic patients. Specifically, Norepinephrine (NE) levels were measured, and CD4+/CD8+ T cells were quantified to assess changes influenced by Esmolol administration. Additionally, cytokine profiles, Procalcitonin (PCT) levels, complete blood counts (CBC), and routine biochemical functions were monitored through data retrieved from EHR systems, providing a broad perspective on patient health and response to treatment. This multifaceted approach aimed to determine how Esmolol affects key immune parameters and overall patient outcomes, addressing both the direct and systemic impacts of this treatment on septic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 90 years.
2. Diagnosed with sepsis or septic shock according to the diagnostic criteria in Suivival Sepsis of 2021.
3. Received adequate fluid resuscitation and necessary exogenous Norepinephrine (NE).
4. No contraindications to Esmolol and appropriate heart rate levels determined by clinical assessment.
5. Provided written informed consent.

Exclusion Criteria:

1. Deceased within three days following ICU admission.
2. Pregnant or lactating individuals.
3. Underwent surgical procedures within the last two weeks.
4. Severe cardiac failure exceeding NYHA Class III.
5. Usage of long-term oral β-blockers or any form of extracorporeal circulation within the last two weeks.
6. Presenting with sinus bradycardia or atrioventricular block.
7. Received high doses of corticosteroids in the past three months.
8. Underwent significant hormone therapy, persistent blood loss of more than 500 ml within any 24-hour period, or were treated with Esmolol for less than three days.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Impact of Esmolol on Survival Rates | Survival rates will be monitored from the time of randomization until the end of the study period or until patient death, whichever comes first, up to 28 days post-randomization.
  The primary outcome measure will be the comparison of survival rates between the treatment and control groups. A logistic regression analysis will be employed to evaluate the effect of Esmolol on survival rates and clinical outcomes, adjusting for potential confounders. Additionally, Kaplan-Meier survival curves will be generated for each group, and a Log-rank test will be used to compare the differences in survival rates over the study period.
Improvement in Organ Function and Inflammatory Markers | Organ function and inflammatory markers will be measured at baseline, then regularly throughout the patient's stay in the ICU, up to a maximum of 28 days.
  As a secondary outcome, the study will assess the effect of Esmolol on organ function and systemic inflammation. This will be evaluated using a composite of changes in organ function scores (such as SOFA - Sequential Organ Failure Assessment score) and levels of inflammatory markers (such as C-reactive protein and IL-6). The analysis will determine if Esmolol correlates with an improvement in these clinical parameters, suggesting a protective or restorative effect on organ function.

SECONDARY OUTCOMES:
Length of Intensive Care Unit (ICU) Stay | From the date of ICU admission until the date of ICU discharge, assessed up to 90 days.
  The duration of ICU stay will be measured to determine if Esmolol administration correlates with a shorter ICU admission period. This measure can reflect the overall impact of the drug on the severity and progression of sepsis, potentially indicating more rapid patient stabilization and recovery.
Reduction in Inflammatory Markers | Baseline and then daily measurements in ICU up to 28 days.
  The study will evaluate the effect of Esmolol on systemic inflammation by measuring changes in inflammatory markers such as C-reactive protein (CRP) and interleukin-6 (IL-6) levels. A decrease in these markers could indicate a beneficial anti-inflammatory effect of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, doctoral, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Result] Pedicino D, Volpe M. beta1-Adrenergic receptor stimulation modulates immune response in cancer: a role for beta-blockers in antineoplastic treatment? Eur Heart J. 2024 Mar 14;45(11):870-871. doi: 10.1093/eurheartj/ehae008. No abstract available. PMID 38240494
- [Derived] Jing D, Xiong L, Zhang R, Fang H, Chen L. Esmolol improves sepsis outcomes through cardiovascular and immune modulation. Front Pharmacol. 2025 May 12;16:1498227. doi: 10.3389/fphar.2025.1498227. eCollection 2025. PMID 40421209

DOCUMENTS (2):
  • Study Protocol (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT06390748/Prot_000.pdf
  • Informed Consent Form (2024-03-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT06390748/ICF_001.pdf